CLINICAL TRIAL: NCT04563520
Title: aPCC and Emicizumab Safety Study in Congenital Hemophilia A Patients With Inhibitors (SAFE Study: Safety of aPCC Following Emicizumab Prophylaxis)
Brief Title: SAFE Study: Safety of aPCC Following Emicizumab Prophylaxis
Acronym: SAFE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Sidonio, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000804; 2025P010684 (Other: Emory IRB)
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hemophilia A
Keywords: hemostatic efficacy; safety; prothrombin complex concentrate
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — emicizumab; anti-inhibitor coagulant complex; recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental treatment (Experimental): Participants will have a first/baseline thrombin generation assay (TGA) sample (to be processed within 60 minutes), followed by an infusion at 15 U/kg dose of aPCC, and provide a second TGA sample 15-30 minutes after to be processed within 60 minutes. If required, a subsequent TGA sample will be obtained upon a 25 U/kg dose of aPCC to be processed within 60-90 minutes.
  Interventions: Drug: Emicizumab; Drug: FEIBA; Drug: rFVIIa

INTERVENTIONS:
Drug: Emicizumab — HEMLIBRA® is a bispecific factor IXa- and factor X-directed antibody indicated for routine prophylaxis to prevent or reduce the frequency of bleeding episodes in adult and pediatric patients ages newborn and older with hemophilia A (congenital factor VIII deficiency) with or without factor VIII inhibitors.
  Other Names: ACE910, Hemlibra and RO5534262
Drug: FEIBA — FEIBA™ is an Anti-Inhibitor Coagulant Complex indicated for use in hemophilia patients with inhibitors for: control and prevention of bleeding episodes, perioperative management, and routine prophylaxis to prevent or reduce the frequency of bleeding episodes.
  The max dose allowed for aPCC will be 50 U/kg dose given at a single visit.
  Other Names: Activated prothrombin complex (aPCC); Anti-Inhibitor Coagulant Complex
Drug: rFVIIa — rFVIIa is a coagulation factor VIIa concentrate indicated for the treatment and control of bleeding episodes occurring in adults and adolescents with hemophilia with inhibitors.
  Other Names: Recombinant activated factor VII

SUMMARY:
The purpose of the aPCC-emicizumab safety study is to investigate the hemostatic efficacy as measured by thrombin generation, of a low personalized dose of aPCC (FEIBA) in children and adults with hemophilia A and inhibitors on emicizumab prophylaxis.

DETAILED DESCRIPTION:
Hemophilia A (HA) is a congenital bleeding disorder caused by deficient or dysfunctional factor VIII (FVIII) which leads to bleeding correlated with factor deficiency severity. Patients with HA develop recurrent bleeds into joints and soft tissues that culminate into debilitating arthropathy and long-term morbidity.

The previous standard of care for high titer antibody eradication in hemophilia A (HA) included a labor-intensive, immune tolerance induction (ITI) regimen administered with concomitant bypassing agent (BPA) prophylaxis, either daily recombinant activated factor VII (rFVIIa) or at least 3 non-consecutive days of activated prothrombin complex concentrate (aPCC) given intravenously (IV) each week.

The overall objective is to determine whether the thrombin generation assay can be used to personalize a dose of aPCC that could be used in a future study during an acute bleeding event and peri-surgical prophylaxis in children and adults with hemophilia A and inhibitors on emicizumab primary prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Moderately severe hemophilia A, defined as FVIII level <0.05 IU/mL before development of an inhibitor
* Age ≥6 years of age at time of informed consent
* Documented on 2 occasions a high titer inhibitor (>5 BU/mL) with a 72-hour washout within 2 years of enrollment
* Parent/guardian (Legally Authorized Representative) or the patient has provided written informed consent
* Adequate hematologic function (Hgb >8 g/dL and platelet count >100,000 µL)
* Adequate hepatic function (total bilirubin ≤1.5 x ULN and both AST/ALT ≤3x ULN at screening (excluding known Gilbert's)
* Adequate renal function (≤2.5 x ULN and CrCl ≥30 mL/min)

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than hemophilia A excluding low VWF (>30% VWF:RCo or VWF:GP1bm)
* Had an active bleed requiring factor therapy at screening
* Previous or current treatment for thromboembolic disease or signs of thromboembolic disease (excluding previously resolved line-associated thrombosis)
* Had a surgical procedure 14 days before screening
* Conditions that may increase the risk of bleeding or thrombosis
* If the patient is treated with rFVIIa or aPCC seven days before screening
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Had current use of any medication other than emicizumab that could affect the coagulation system.
* Known HIV infection with CD4 count <200 cells/µL within 24 weeks before screening. Testing is not required if <35 years of age.
* Use of systemic immunomodulators at enrollment or planned use during the study
* Participants who are at high risk for TMA (for example, have a previous medical/family history of TMA), in the investigator's judgment
* Concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study, may pose an additional risk, or would, in the opinion of the investigator, preclude the participant's safe participation in and completion of the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Thrombin generation capacity after aPCC (FEIBA) infusion | Baseline and up to 30 minutes after infusion
  Thrombin generation capacity from up to two escalating doses of aPCC will be measured using a thrombin generation assay at baseline and up to 30 minutes after FEIBA infusion.

SECONDARY OUTCOMES:
Number of serious adverse events | up to 1 year
  Number of serious adverse events will be recorded
Number of serious bleeding episodes | up to 1 year
  Number of serious bleeding episodes will be recorded
Number of episodes of thrombotic events including thrombotic microangiopathy (TMA) | up to 1 year
  Number of episodes of thrombotic events including thrombotic microangiopathy (TMA) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sidonio, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification, will be available
Supporting Information: Study Protocol, SAP, ICF